CLINICAL TRIAL: NCT00195728
Title: An Open-Label Study Evaluating the Safety and Tolerability of Long Term Administration of Hydrocodone/Acetaminophen Extended ReleaseTablets (Vicodin® CR) in Subjects With Moderate to Severe Chronic, Non-Malignant Pain
Brief Title: Long Term Safety and Tolerability Study in Approximately 350 Subjects With Moderate to Severe Chronic, Non-malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Andrea Best, DO, MPH, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M03-666
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Moderate to Severe Chronic, Non-malignant Pain
Keywords: Hydrocodone/Acetaminophen; Vicodin CR
MeSH Terms: interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: Hydrocodone/Acetaminophen on Extended Release

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen on Extended Release — 2 tablets twice daily
  Other Names: ABT-712

SUMMARY:
The purpose of the study is to evaluate the safety of Vicodin CR (combination opioid and acetaminophen containing product) in patients with chronic pain due to osteoarthritis or low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between 21 and 75 years of age

  * Females must be of non-child bearing potential or practicing birth control
* Moderate to severe mechanical low back pain OR moderate to severe OA of the hip or knee pain
* Require medicine for pain the majority of days in the previous 3 months, AND for at least 4 days per week, during the previous 4 weeks.
* Pain is not controlled with non-opioid analgesics or is contraindicated due to side effects and/or currently receiving opioid therapy equivalent to 40 mg/day of morphine or less

Exclusion Criteria:

* Pregnant and/or breastfeeding females or females planning to become pregnant during the course of the study
* Incapacitated, bedridden, or confined to a wheelchair permitting little or no self-care
* Injury to the index joint or lower back within 3 months of study
* History of any of the following:

  * Major surgery to the lower back within the last 5 years OR
  * Joint replacement/reconstruction to the index joint OR
  * Arthroscopic or open surgery to the index joint within the last year OR
  * Any surgery within 3 months of study
* Osteoporotic compression fracture, traumatic vertebral fracture or invasive intervention for low back pain within the last year.
* Abnormal neurological exam, or lower extremity symptoms characteristic of neurogenic pain
* History of inflammatory or infectious arthritis, tumors or infections of spinal cord, spinal stenosis, fibromyalgia or other chronic painful condition
* Severe gastrointestinal narrowing
* History of peritonitis, cystic fibrosis, chronic intestinal eudoobstruction, or Meckel's diverticulum.
* Has received

  * Oral, intramuscular (IM), intravenous (IV) or non-index joint intra- articular corticosteroids within 1 month of study OR
  * Intra-articular corticosteroids at the index joint or epidural corticosteroids to the lower back region within 2 months of study, OR
  * Viscosupplementation therapy to index joint within 4 months of study
* History of drug (licit or illicit) or alcohol abuse/addiction
* Positive result for drugs of abuse at screening.
* Chronic heavy drinker, consuming more than 4 alcoholic drinks per day.
* History of malnutrition or starvation or is likely to fast for more than 4 consecutive days during the course of the study.
* Medical condition or illness other than OA/CLBP, which is not well controlled
* History of allergic reaction or a clinically significant sensitivity or intolerance to opioids and/or acetaminophen.
* Newly diagnosed medical condition
* Clinically significant infection/injury/illness within 1 month of study
* Receiving systemic chemotherapy, or has an active malignancy of any type, or has been diagnosed with cancer within the past 5 years. Basal cell carcinoma of the skin that has been successfully treated will be permitted.
* Known or suspected history of Human Immunodeficiency Virus.
* Positive Hepatitis Screen
* Clinically significant abnormalities in clinical chemistry, hematology or urinalysis
* Received any investigational drug within 1 month of study
* History of major psychiatric disorder
* Active or uncontrolled seizure disorder.
* Requires treatment with monoamine oxidase inhibitors (MAOIs), or tricyclic antidepressants during the course of the study.
* Surgical procedure planned, or scheduled during the course of this study.
* Ongoing workman's compensation claim or litigation.
* Previous participation in the M03-666 study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety evaluation | 56 weeks
  Long term safety

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — Abbott
Locations (76):
- United States (76):
  - Site Ref # / Investigator 1696, Huntsville, Alabama
  - Site Reference # / Investigator 1729, Chandler, Arizona
  - Site Reference # / Investigator 1702, Mesa, Arizona
  - Site Reference # / Investigator 1745, Peoria, Arizona
  - Site Ref # / Investigator 1697, Tempe, Arizona
  - Site Ref # / Investigator 1818, Tempe, Arizona
  - Site Reference # / Investigator 1795, Tucson, Arizona
  - Site Ref # / Investigator 2555, Carmichael, California
  - Site Reference # / Investigator 1688, Fair Oaks, California
  - Site Reference # / Investigator 1790, Pasadena, California
  - Site Reference # / Investigator 1735, San Diego, California
  - Site Reference # / Investigator 1775, San Luis Obispo, California
  - Site Ref # / Investigator 1742, Santa Ana, California
  - Site Ref # / Investigator 1754, Tarzana, California
  - Site Reference # / Investigator 1700, Whittier, California
  - Site Reference # / Investigator 1690, Colorado Springs, Colorado
  - Site Ref # / Investigator 1713, Littleton, Colorado
  - Site Ref # / Investigator 1711, Bristol, Connecticut
  - Site Reference # / Investigator 1723, Clearwater, Florida
  - Site Ref # / Investigator 1813, Clearwater, Florida
  - Site Reference # / Investigator 1718, DeLand, Florida
  - Site Reference # / Investigator 1819, Longwood, Florida
  - Site Reference # / Investigator 1809, Miami, Florida
  - Site Reference # / Investigator 1738, Miami, Florida
  - Site Ref # / Investigator 1716, Orlando, Florida
  - Site Reference # / Investigator 1755, Palm Harbor, Florida
  - Site Ref # / Investigator 1814, Pembroke Pines, Florida
  - Site Reference # / Investigator 1737, Plantation, Florida
  - Site Reference # / Investigator 1747, St. Petersburg, Florida
  - Site Reference # / Investigator 1744, Arlington Heights, Illinois
  - Site Reference # / Investigator 1691, Chicago, Illinois
  - Site Reference # / Investigator 1714, Evansville, Indiana
  - Site Ref # / Investigator 1739, Metairie, Louisiana
  - Site Reference # / Investigator 1810, Owings Mills, Maryland
  - Site Ref # / Investigator 1707, Fall River, Massachusetts
  - Site Reference # / Investigator 1743, Wellesley Hills, Massachusetts
  - Site Ref # / Investigator 1792, Jackson, Mississippi
  - Site Reference # / Investigator 1721, St Louis, Missouri
  - Site Ref # / Investigator 1812, St Louis, Missouri
  - Site Reference # / Investigator 2424, St Louis, Missouri
  - Site Ref # / Investigator 1722, Omaha, Nebraska
  - Site Ref # / Investigator 1774, Omaha, Nebraska
  - Site Reference # / Investigator 1789, Omaha, Nebraska
  - Site Reference # / Investigator 1705, Las Vegas, Nevada
  - Site Reference # / Investigator 1791, Las Vegas, Nevada
  - Site Reference # / Investigator 1701, Medford, New Jersey
  - Site Reference # / Investigator 2461, Trenton, New Jersey
  - Site Reference # / Investigator 1726, Binghamton, New York
  - Site Reference # / Investigator 1815, New York, New York
  - Site Reference # / Investigator 1708, Charlotte, North Carolina
  - Site Ref # / Investigator 1730, Monroe, North Carolina
  - Site Reference # / Investigator 1741, Raleigh, North Carolina
  - Site Reference # / Investigator 1689, Cincinnati, Ohio
  - Site Ref # / Investigator 1694, Cincinnati, Ohio
  - Site Ref # / Investigator 1816, Cleveland, Ohio
  - Site Reference # / Investigator 1715, Oklahoma City, Oklahoma
  - Site Reference # / Investigator 2423, Portland, Oregon
  - Site Reference # / Investigator 1794, Beaver, Pennsylvania
  - Site Reference # / Investigator 1749, Duncansville, Pennsylvania
  - Site Reference # / Investigator 1752, Erie, Pennsylvania
  - Site Reference # / Investigator 1709, Mechanicsburg, Pennsylvania
  - Site Reference # / Investigator 1757, Cordova, Tennessee
  - Site Reference # / Investigator 1727, Selmer, Tennessee
  - Site Ref # / Investigator 1692, Austin, Texas
  - Site Reference # / Investigator 1722, Austin, Texas
  - Site Reference # / Investigator 2425, Dallas, Texas
  - Site Reference # / Investigator 1699, Fort Worth, Texas
  - Site Ref # / Investigator 1725, Killeen, Texas
  - Site Reference # / Investigator 1710, San Angelo, Texas
  - Site Reference # / Investigator 1686, San Antonio, Texas
  - Site Reference # / Investigator 2426, San Antonio, Texas
  - Site Reference # / Investigator 1808, San Antonio, Texas
  - Site Reference # / Investigator 1732, Salt Lake City, Utah
  - Site Reference # / Investigator 1740, Salt Lake City, Utah
  - Site Ref # / Investigator 1733, Norfolk, Virginia
  - Site Reference # / Investigator 1719, Virginia Beach, Virginia